CLINICAL TRIAL: NCT00291369
Title: PERCY QUATTRO: Medroxyprogesterone, Interferon Alpha-2a, Interleukin 2 or Combination of Both Cytokines in Patients With Metastatic Renal Carcinoma of Intermediate Prognosis
Brief Title: Cytokines in Patients With Metastatic Renal Cell Carcinoma of Intermediate Prognosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: French Immunotherapy Intergroup (Other); SCAPP (Sub-Cutaneous Administration Proleukin Program) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERCY QUATTRO; ET99-058
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2006-02

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic renal cell carcinoma; Interleukin-2; Interferon alfa; Cytokines; Survival
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interleukin-2; Interferon-alpha; Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Interleukin-2
Drug: Interferon alfa
Drug: medroxyprogesterone acetate

SUMMARY:
The PERCY Quattro trial has been designed to evaluate the survival benefit of two cytokine treatments, Interleukin-2 (IL2) and/or alpha interferon (IFN), for patients with intermediate chance of response in metastatic renal cell carcinoma.

Eligible patients will be randomly assigned in a two-by-two factorial design to either medroxyprogesterone (MPA), subcutaneous IFN, subcutaneous IL2, or a combination of IFN and IL2.

The primary objective of the study is overall survival; secondary objectives are progression-free survival, response rate, toxicity, and quality of life.

DETAILED DESCRIPTION:
The PERCY Quattro trial has been designed to evaluate the survival benefit of Interleukin-2 (IL2) and/or alpha interferon (IFN) for patients with intermediate chance of response in metastatic renal cell carcinoma.

The primary objective is overall survival, and secondary objectives are progression-free survival, response rate, toxicity, and quality of life assessed before and after induction treatment (week 10).

Patients above 18 years of age are eligible if they have histologically confirmed, clearly progressive metastatic renal carcinoma, more than one metastatic organ and good performance status (Karnofsky score ≥80%), or one metastatic organ with Karnofsky score 80%, normal blood and liver functions with creatinine level <= 160 µmol/L.

Eligible patients will be randomly assigned in a two-by-two factorial design to either medroxyprogesterone (MPA), subcutaneous IFN, subcutaneous IL2, or a combination of IFN and IL2. The planned sample size is 456 patients (114 in each of the four arms). MPA is given orally as 200 mg daily. IFN is given subcutaneously as 9 million IU three times a week. IL2 is given subcutaneously on a four-week schedule: 9 million IU twice daily for five days followed by a two-day rest, then, on the following three weeks, 9 million IU twice daily for two days then 9 million IU once daily on the following three days; after a week of rest, an identical 4-week cycle is administered. IFN and IL2 combination is given using identical routes, schedules and doses except for a reduction of IFN dose to 6 million IU per injection.

ELIGIBILITY:
Inclusion Criteria:

* Progressive histologically proven metastatic renal cell carcinoma.
* Patient with only 1 metastatic site and Karnofsky = 80% or more than 1 metastatic site and Karnofsky >= 80%.
* Age >= 18
* No wide-field radiation therapy for 6 weeks at least.
* No active brain metastasis.
* Blood values within limits of normal (hematocrit > 30% and leukocyte count >= 4x109/l and platelet count >= 120x109/l).
* Creatinine < 150 µmol/l and bilirubin <= normal.
* Female patients of childbearing potential: effective method of contraception is necessary.
* Written, voluntary, informed consent.

Exclusion Criteria:

* Previous treatment with cytokines.
* Only one metastatic organ and Karnofsky = 90% or 100% (inclusion in good prognosis group).
* More than one metastatic organ (at least one metastasis to the liver) and <12 months between initial diagnosis and diagnosis of metastasis.
* Active brain metastases.
* Patient with concurrent grade III/IV heart disorder (congestive heart failure, coronary artery disease, uncontrolled hypertension, severe arrhythmia, etc) and/or stroke volume < 50%.
* Severe pulmonary, hepatic, or renal disease potentially aggravated by treatment.
* Severe concurrent infection necessitating antibiotics
* Patient with known HIV or AIDS-related disease, or presence of HB antigen or known chronic hepatitis.
* Previous allograft.
* Patient under corticosteroid treatment.
* Previous or concurrent primary malignancies at other sites (except from baso-cellular skin cancer or cervical cancer in situ)
* Pregnant or lactating woman.
* Follow-up difficult because of geography or personal circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456
Dates: Start 1999-12; Study Completion 2005-02

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival
Objective response rate
Toxicity
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Negrier, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

REFERENCES:
- [Background] Negrier S, Escudier B, Lasset C, Douillard JY, Savary J, Chevreau C, Ravaud A, Mercatello A, Peny J, Mousseau M, Philip T, Tursz T. Recombinant human interleukin-2, recombinant human interferon alfa-2a, or both in metastatic renal-cell carcinoma. Groupe Francais d'Immunotherapie. N Engl J Med. 1998 Apr 30;338(18):1272-8. doi: 10.1056/NEJM199804303381805. PMID 9562581
- [Background] Ravaud A, Delva R, Gomez F, Chevreau C, Douillard JY, Peny J, Coudert B, Negrier S; Groupe Francais d'Immunotherapie. Subcutaneous interleukin-2 and interferon alpha in the treatment of patients with metastatic renal cell carcinoma-Less efficacy compared with intravenous interleukin-2 and interferon alpha. Results of a multicenter Phase II trial from the Groupe Francais d'Immunotherapie. Cancer. 2002 Dec 1;95(11):2324-30. doi: 10.1002/cncr.10968. PMID 12436438
- [Background] Negrier S, Escudier B, Gomez F, Douillard JY, Ravaud A, Chevreau C, Buclon M, Perol D, Lasset C. Prognostic factors of survival and rapid progression in 782 patients with metastatic renal carcinomas treated by cytokines: a report from the Groupe Francais d'Immunotherapie. Ann Oncol. 2002 Sep;13(9):1460-8. doi: 10.1093/annonc/mdf257. PMID 12196373